CLINICAL TRIAL: NCT03280732
Title: Lung Ultrasound in Diagnosing and Monitoring of Pulmonary Complications in Children With Acute Bronchiolitis
Brief Title: Use of Lung Ultrasound in Children With Acute Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Marcello Lanari, Director, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/2016/O/Sper
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Bronchiolitis Acute
Keywords: Lung Ultrasound; Chest X-Ray; Pneumonia; Pneumothorax; Pleural effusion
MeSH Terms: conditions — Pneumonia; Pneumothorax; Pleural Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Ultrasound (Experimental): Bedside lung ultrasound will be performed by a paediatrician with specific LUS expertise and blinded to clinical and radiological data.
  Interventions: Device: Lung Ultrasound

INTERVENTIONS:
Device: Lung Ultrasound — A Mindray-DC-T6 ultrasound machine equipped with a linear probe with frequencies ranging from 7.5 to 12 MHz will be use. LUS examination will consist of both longitudinal and transversal sections according to the methodology described by Copetti and colleagues.

SUMMARY:
Bronchiolitis is the leading cause of hospitalization in infants. The diagnosis is clinical and chest x-ray (CXR) should be reserved for severe cases in which signs of pulmonary complications are present. Nevertheless, CXR is performed in more than 50% of hospitalized patients with bronchiolitis, which exposes infants to ionizing radiation.

Data on the possible role of lung ultrasound (LUS) in children with bronchiolitis and suspected pulmonary complications have not been published yet.

The purpose of this study is to evaluate the use of LUS compared to CXR in diagnosing and monitoring pulmonary complications (pneumonia, pleural effusion, pneumothorax) in children with acute bronchiolitis. The second purpose of the study is to evaluate the correlation between clinical course and ultrasound findings in children with bronchiolitis.

The inclusion of LUS in the diagnostic work-up of bronchiolitis could possibly reduce the misuse of CXR in infants and the exposure to ionizing radiations.

DETAILED DESCRIPTION:
Bronchiolitis is the most common lower respiratory tract infection that affects children younger than 24 months. The diagnosis is clinical and, according to international guidelines, chest x-ray (CXR) should be reserved for cases in which signs of pulmonary complications are present or where respiratory effort is severe to warrant intensive care unit admission. Despite these recommendations, CXR is still performed in about 50% of bronchiolitis (ranging from 24 to 77%), which exposes infants to ionizing radiation.

Given its portability, no ionizing radiation, rapid and repeat testing, lung ultrasound (LUS) has become an emerging diagnostic tool for pneumonia, pleural effusion and pneumothorax in adults and children. At present, LUS is not included in the diagnostic work-up of bronchiolitis. Previous papers have reported that LUS may be useful in bronchiolitis because of a good correlation between clinical course and ultrasound findings. However, data on the possible role of LUS in children with bronchiolitis and suspected pulmonary complications have not been published yet.

Enrolled patients will undergo a bedside LUS in the first 12 hours after CXR. LUS will be performed by one paediatrician with specific LUS expertise and blinded to clinical and radiological data. The paediatrician must have previously attended a specific course on LUS and supervised practical training. A Mindray-DC-T6 ultrasound machine equipped with a linear probe with frequencies ranging from 7.5 to 12 MHz will be use. LUS examination will consist of both longitudinal and transversal sections from the anterior, lateral and posterior chest wall according to the methodology described by Copetti et al. A radiologist will then independently repeat the LUS to test the sonographer inter-observer agreement. The radiologist will be blinded to the results of the previous studies (LUS and CXR). The LUS findings will be recorded on the data form together with patient demographics, symptoms, CXR findings and laboratory data.

Patients with LUS positive for pulmonary complications will receive follow-up ultrasound every 48 hours until the resolution or the discharge.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized with a diagnosis of bronchiolitis
* Age < 24 months
* CXR as part of usual clinical practice because of clinical suspicion of pulmonary complications
* Informed written consent

Exclusion Criteria:

* chronic respiratory disease (i.e. bronchopulmonary dysplasia)
* congenital heart disease
* severe neuromuscular disease
* congenital or acquired immunodeficiency

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
LUS vs CXR in diagnosing pulmonary complications in bronchiolitis | 12 hours
  To evaluate the use of LUS compared to CXR to diagnose pulmonary complications (pneumonia, pleural effusion, pneumothorax) in children with acute bronchiolitis

SECONDARY OUTCOMES:
Sonographer inter-observer agreement | 12 hours
  To evaluate the sonographer inter-observer agreement between a paediatrician and a paediatric radiologist in the diagnosing of pulmonary complications in children with acute bronchiolitis
LUS and severity of bronchiolitis | 12 hours
  - To evaluate the correlation between clinical course and ultrasound findings in children with bronchiolitis.

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Lanari, Professor, Principal Investigator — Pediatric Emergency Unit, S. Orsola-Malpighi Hospital, University of Bologna
Locations (1):
- Pediatric Emergency Unit, S. Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Background] Parikh K, Hall M, Mittal V, Montalbano A, Mussman GM, Morse RB, Hain P, Wilson KM, Shah SS. Establishing benchmarks for the hospitalized care of children with asthma, bronchiolitis, and pneumonia. Pediatrics. 2014 Sep;134(3):555-62. doi: 10.1542/peds.2014-1052. PMID 25136044
- [Background] Florin TA, Byczkowski T, Ruddy RM, Zorc JJ, Test M, Shah SS. Variation in the management of infants hospitalized for bronchiolitis persists after the 2006 American Academy of Pediatrics bronchiolitis guidelines. J Pediatr. 2014 Oct;165(4):786-92.e1. doi: 10.1016/j.jpeds.2014.05.057. Epub 2014 Jul 9. PMID 25015578
- [Background] Mazrani W, McHugh K, Marsden PJ. The radiation burden of radiological investigations. Arch Dis Child. 2007 Dec;92(12):1127-31. doi: 10.1136/adc.2006.101782. PMID 18032642
- [Background] Copetti R, Cattarossi L. Ultrasound diagnosis of pneumonia in children. Radiol Med. 2008 Mar;113(2):190-8. doi: 10.1007/s11547-008-0247-8. Epub 2008 Apr 2. English, Italian. PMID 18386121
- [Derived] Biagi C, Pierantoni L, Baldazzi M, Greco L, Dormi A, Dondi A, Faldella G, Lanari M. Lung ultrasound for the diagnosis of pneumonia in children with acute bronchiolitis. BMC Pulm Med. 2018 Dec 7;18(1):191. doi: 10.1186/s12890-018-0750-1. PMID 30526548